CLINICAL TRIAL: NCT01064960
Title: Clinical Trial Protocol for Therapeutic MRI-guided High Intensity Focused Ultrasound Ablation of Uterine Fibroids in a 3T MRI Scanner
Brief Title: Therapeutic MRI-HIFU Ablation of Uterine Fibroids in a 3T MRI Scanner
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 997677
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Uterine Leiomyomas
Keywords: Neoplasms, Connective and Soft Tissue; Neoplasms, Muscle Tissue; Neoplasms; Myofibroma; Neoplasms by Histologic Type; Connective Tissue Diseases; Neoplasms, Connective Tissue; Leiomyoma
MeSH Terms: conditions — Myofibroma; Neoplasms, Connective and Soft Tissue; Neoplasms, Muscle Tissue; Neoplasms; Neoplasms by Histologic Type; Connective Tissue Diseases; Neoplasms, Connective Tissue; Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated leiomyomas (Experimental): Pre- or peri-menopausal women with symptomatic uterine fibroids who desire a uterine sparing procedure are treated with the Philips MR-guided HIFU system. Patients must have completed child bearing prior to enrolling in this study.
  Interventions: Device: Philips MR-guided HIFU system

INTERVENTIONS:
Device: Philips MR-guided HIFU system — HIFU is the use of focused ultrasound energy to penetrate through soft tissue and causes localized high temperatures (55°C to 70°C) for a few seconds within the target producing well defined regions of protein denaturation, irreversible cell damage, and coagulative necrosis.
  Other Names: Sonalleve; Uterine Leiomyomas; Fibroids; HIFU; Ablation; High Intensity Focused Ultrasound

SUMMARY:
This study is to collect supplementary safety and technical effectiveness data of Philips MRI guided High Intensity Focused Ultrasound (HIFU) in ablating uterine tissue associated with symptomatic fibroids in a 3T MRI scanner. The importance of this therapy is that it offers a non-invasive, uterine sparing procedure for the treatment of uterine fibroids in pre- and peri- menopausal women. MRI guided high intensity focused ultrasound uses ultrasound to heat and thermally ablate fibroid tissue. The MRI system identifies the ultrasound path and monitors heat rise in the fibroid tissue. The goal of the study is to collect supplementary 3T treatment safety and technical effectiveness data in a 1 month follow-up study. MRguided HIFU will be performed in patients who pass inclusion/exclusion criteria. Safety, quality of life, and imaging endpoints will be evaluated in all study patients.

DETAILED DESCRIPTION:
Fibroids occur in 20-50% of women over 30 years of age, and with increasing size produce pain, menorrhagia, pressure, bloating and urinary and bowel compression symptoms. Fibroids may also cause infertility. Uterine leiomyomas are benign tumors originating from smooth muscle cells of the uterus and occasionally the smooth muscle of uterine blood vessels. Fibroids are estrogen dependent tumors ranging in size and number and can be found within the myometrium(intramural), at the uterine periphery extending to the serosa (subserosal), or pushing into the uterine cavity (submucosal). Symptomatic fibroids impact health and well-being of the female including lost work hours and reduced quality of life.

Current medical treatments include invasive removal of the fibroid (hysterectomy, myomectomy), drug therapy (GnRH analogues or progestin compounds) or treatments causing necrosis of the fibroid tissue such as ablation (freezing or heating) or embolization. For the relief of symptoms, women wishing to preserve the uterus may choose between invasive procedures of myomectomy, Uterine Artery Embolization (UAE), ablation or cryotherapy. The surgically invasive procedures require anesthesia, hospital stays, and long recovery periods. HIFU may offer an alternative to the above mentioned surgically invasive procedures.

In MRI-guided High Intensity Focused Ultrasound (HIFU), the ultrasound generated by the transducer is focused into a small focal tissue volume at specific target locations. During treatment, the beam of focused ultrasound energy penetrates through soft tissue and causes localized high temperatures (55°C to 70°C) for a few seconds within the target producing well defined regions of protein denaturation, irreversible cell damage, and coagulative necrosis. The MRI system allows 3D planning, means of measuring the temperature increase generated by HIFU, and the capability to quantifying the energy/dose delivered to the treatment zone.

This study is a single-center, single arm, non-randomized trial evaluating the safety, technical effectiveness and volume treatment capabilities of the Philips MR-guided HIFU system in the treatment of symptomatic uterine fibroid patients. Patients who have symptomatic uterine fibroids, who are eligible according to the inclusion and exclusion criteria and provide informed consent will be enrolled in this study. It is anticipated that women will participate in the study for a 2month period to include the screening, HIFU treatment and post treatment follow-up.

This clinical study is designed to confirm safety and demonstrate technical effectiveness of the Philips HIFU system for Uterine Fibroid treatment. Safety will be primarily assessed by evaluating minor complications and adverse events, and technical effectiveness will primarily be assessed with MRI measurements. Specific primary and secondary endpoints are detailed below.

The study will use a combination of three primary endpoints: MR imaging of ablated volumes and minor complications/adverse events analysis to establish the safety and technical effectiveness of the Philips MR-HIFU system. These endpoints will determine the trial success.

The treatment capabilities and technical effectiveness of the Philips MR-guided HIFU system will be assessed by (measurement type is noted in parentheses)

1. Comparing the actual MR-measured ablated volumes to MR thermal dose predicted volumes Safety of the Philips MR-guided HIFU system will be demonstrated by
2. Evaluating any minor complications or adverse events that result from the MR-guided HIFU treatment
3. Verifying with MR imaging that no unintended lesions are formed as a result of the Treatment

   In addition, the following endpoints will be collected to supplement the primary outcomes:
4. Pain and discomfort scores before, during and after treatment: These endpoints will be recorded using a 10-point visual analog scale for pain 4-point scale for discomfort.
5. Return to Activity: This duration in days will be determined by the time after which the patients return to work (i.e. days after leaving the hospital) or to the usual activities for those not employed.
6. Length of Hospital Stay (LOS): This duration in hours will be measured from the time the patient will arrive to the hospital until she will leave the hospital.
7. Quality of Life questionnaires: the SF-36(http://www.sf36.org/tools/SF36.shtml) and UFS-QoL (which includes SSS)

ELIGIBILITY:
Inclusion Criteria:

* Women, age between 18 and 59 years
* Weight < 140kg
* Pre- or peri-menopausal
* Uterine size < 24 weeks
* Transformed SSS score > 40
* Normal Cervical cell assessment by PAP
* Symptomatic Fibroid disease
* Dominant fibroid greater than or equal to 3cm and less than or equal to 12 cm

Exclusion Criteria:

* Other Pelvic Disease
* Desire for future pregnancy
* Significant systemic disease even if controlled
* Positive pregnancy test
* Hematocrit < 25%
* Scarring or other interference of the HIFU beam
* MRI or contrast contraindicated
* Fibroids not quantifiable on MRI
* Calcifications around or throughout uterine tissues
* Communication barrier

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety of HIFU for treatment of the uterine fibroids as determined by adverse event reporting. | 30 days after treatment
  Number of adverse events reported in the study divided by the total number of treated subjects.
Technical efficacy of HIFU for treatment of uterine fibroids as assessed by a change in the Symptom Severity Score | 30 days after treatment
  Mean absolute change in the Symptom Severity Score (SSS) of the uterine Fibroid Symptoms Quality of Life questionnaire from baseline to 30 days after treatment.

SECONDARY OUTCOMES:
Change in Quality of Life Scores | 30 days after treatment
  Mean absolute score change in the Quality of Life questionnaire from baseline to 30 days after treatment.
Pain score | 72 hours after treatment
  Mean Visual Analog Score (VAS) for pain 72 hours after treatment.
Timeframe before returning to daily activities | 72 hours after treatment
  Mean timeframe for the patient to return to normal activity after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, Professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511